CLINICAL TRIAL: NCT04355091
Title: Effect of Emotional Freedom Techniques (EFT) on Postpartum Depression
Brief Title: Emotional Freedom Techniques (EFT) and Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Neriman Guducu, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99984023-302.99-
Record Dates: First submitted 2020-04-06; First posted 2020-04-21 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; pregnancy; stress
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: In order to determine the risk of depression, the Edinburgh Postpartum Depression Scale (EPDS) will be administered to the pregnant women. Pregnant women who receive 12 ≥ points from the EPDS will be included in the randomization process.
  Subsequently, the tests will be applied to experimental and control groups. EFT will be applied to women in the experimental group. One or two weeks after the application, it will be discussed again and questioned how she feels, whether that problem still disturbs her. The number of EFT sessions can be increased or decreased depending on the condition of the woman (the average number of sessions reported in the studies ranges from 2-10). After all EFT sessions are completed, three months and six months after the last application, post-tests will be done. the control group will receive routine midwifery care. The post-tests will be done by the control group after three months and six months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The pregnant women in this group will be informed about the application of EFT with a written material.
  The pregnant women who have undergone EFT will be interviewed a week or two after the application, and how they feel and whether the problem still disturbs him. If a new issue is reported, similar actions will be repeated for this new issue. The number of EFT sessions was decided based on the condition of the pregnant woman. After all EFT sessions are completed, a re-evaluation (post-test) of Edinburgh Postpartum Depression Scale, Stress Coping Scale and State-Trait Anxiety Inventory will be done.
  The same participants will be asked to apply the other inventories and the postpartum interview form if she had birth three months and six months after the last application (follow-up). In the follow-up study performed three months after the last application, EFT will be applied to the pregnant women in need.
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- control group (No Intervention): The participants in this group will be talked about the problems they should have in routine midwifery care, the problems they encounter during pregnancy or postpartum period and the subjects they want to receive information.
  If necessary, suggestions will be made for problems related to pregnancy, postpartum period or newborn care. Again, with these participants, after the depression risk determination (pre-test), after the interviews ended (post-test), three months and six months after the last application, Edinburgh Postpar All Depression Scale, Stressful Life Events List, Stress Coping Scale. If the pregnant woman has given birth, State-Trait Anxiety Inventory and postnatal interview form will be performed.

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT) — It combines cognitive therapy, acceptance and stability therapy, and acupuncture point stimulation, and is based on manual stimulation of acupuncture points specific to Shiatsu or other acupressure massage forms, rather than using acupuncture needles.
  Arms: Intervention Group

SUMMARY:
Hypothesis 1: Pregnant women in the EFT group will have a lower test score from Edinburgh Postpartum Depression Scale, and a follow-up score of three months and six months after the last application date, compared to the control group.

Hypothesis 2: In the post-test of pregnant women in the EFT group, three months and six months after the last application date, the optimistic, self-confident and social support approach methods used to deal with stress will increase, and the helpless and submissive approach styles will decrease compared to the control group.

Hypothesis 3: Pregnant women in the EFT group will have a lower test score from the State-Trait Anxiety Inventory, and a follow-up score of three months and six months after the last application date, compared to the control group.

DETAILED DESCRIPTION:
In addition to being a natural life event for women, pregnancy is also a period in which significant biological and psychosocial changes are experienced, and the risk of encountering many factors that may create anxiety and stress. While many women easily adapt to these changes occurring with pregnancy and childbirth, some women may develop various levels of mental illness. It is reported that the majority of depression, one of the mental illnesses, occurs in women aged 18-44, including fertility processes such as pregnancy, childbirth, and puerperium. A meta-analysis on the subject indicates that the rate of depression increases in pregnancy and postpartum period.

Depression during pregnancy can cause serious effects for all family members. Pregnancy depression which is not managed well, damages the developing fetüs due to problems such as poorly managed pregnancy depression, substance abuse, insufficient prenatal care, and suicide attempt. It also causes an increased level of cortisol, which can lead to insulin resistance and, if not compensated, gestational diabetes may occur. In this process, elevated norepinephrine and cortisol reduce blood flow to the uterus, causing very serious obstetric and neonatal consequences both on pregnant and fetus, and pregnancy-related adverse events such as HT and preeclampsia are also increasing. Postpartum depression is the most negative result of untreated depression during pregnancy.

In the initial treatment of pregnancy depression and postpartum depression, good psychosocial evaluation, activation of support systems and the combined use of integrated therapies are the most ideal options. Treatment options for postpartum depression are psychotherapy (interpersonal relationships therapy and cognitive - behavioral therapy), drug therapy and non-pharmacology applications. While it is recommended to apply psychotherapy and non-pharmacological approaches as the first choice in mild depression, the use of pharmacological treatments (antidepressants) stands out in moderate and severe depression.

One of the psychotherapeutic techniques, whose numbers have increased rapidly in recent years, is "Emotional Freedom Techniques (EFT)". EFT; It combines cognitive therapy, acceptance and stability therapy, and acupuncture point stimulation, and is based on manual stimulation of acupuncture points specific to Shiatsu or other acupressure massage forms, rather than using acupuncture needles.Manual pressure on acupuncture sites has been found to be as effective as acupuncture needling technique.It is an initiative that can be applied by individuals and midwives easily after receiving the necessary education all over the world.

EFT has a comprehensive research bibliography that includes successful treatment of various psychological conditions such as depression, anxiety, phobias, and post-traumatic stress disorder. The duration of treatment in these studies varies from one to ten sessions. Feinstein states that in EFT studies that include a follow-up assessment, participants maintain their profit and the rehabilitation period varies between 3 months and 2 years.

Considering all these data, it is necessary to focus primarily on the prenatal period in order to develop preventive and therapeutic interventions. In the literature, scientific studies evaluating the effectiveness of EFT on depression are included, but only one study has been reached in which EFT is applied during pregnancy, and this study is related to stress and endurance. In addition, with this study, an important step will be taken to include an easy-to-apply, inexpensive therapeutic method such as pregnancy and postpartum depression treatments, and evidence will be sought to ensure that all professionals dealing with women's health, especially midwifery, use this technique.

The aim of the study is to evaluate the effect of EFT on postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* To be in the 18-49 age range
* To be at least a primary school graduate
* To be pregnant between 13-30 weeks
* Not having a risky pregnancy,
* Having spontaneous pregnancy,
* Having a single and live fetus
* Not having a chronic serious physical illness or disability
* The absence of infection, wound, scar in the tapping area

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 140 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Edinburgh Postpartum Depression Scale scores at 6 months | Baseline and 6 months
  The scale consists of 10 items. Items are evaluated in 4-point Likert format and scored between 0-3. The lowest score that can be obtained from the scale is 0, the highest score is 30. Each item is scored as 0,1,2,3 in the scale.
  In the evaluation of 3,5,6,7,8,9,10 items, the scoring is reversed (3,2,1,0). Individuals with a total scale score higher than the cut-off point are considered a risk group for depression. The cut-off score was taken as 12 in this study.

SECONDARY OUTCOMES:
Stress Coping Styles Scale | Change from baseline in stress coping styles at 6 months
  This scale is used to determine the coping mechanisms used by the participants in the face of stressful situations.It consists of 30 items and 5 sub-dimensions.
  High scores from each of the five subscales identified indicate an increase in the use of coping style expressed by that subscale. These subscales and the items are as follows:
  1. Self-Confident Approach: 8, 10, 14, 16, 20, 23, 26,
  2. Optimistic Approach: 2, 4, 6, 12 18,,
  3. Helpless Approach: 3, 7, 11, 19, 22, 25, 27, 28,
  4. Submissive Approach: 5, 13, 15, 17, 21, 24,
  5. Contacting Social Support: 1, 9, 29, 30. Items 1 and 9 in the scale are reversed. Subgroup scores are obtained by dividing the score from each sub-dimension by the number of items.
State-Trait Anxiety Inventory | Change from baseline in State-Trait Anxiety scores at 6 months
  This scale consists of a total of forty items; the "State Anxiety Scale" consisting of twenty items and the "Trait Anxiety Scale" consisting of twenty items. There are two types of expressions in the scales: direct and reversed. Direct expressions express negative emotions, and reversed expressions express positive emotions. There are ten (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20th) reversed statements on the state anxiety scale. On the trait anxiety scale, there are seven (1, 6, 7, 10, 13, 16, 19th items) reversed. The total score value obtained from each scale is between minimum 20 and maximum 80. The total score of the reverse expressions is subtracted from the total score obtained for direct expressions. A predetermined and constant value is added to this number. This is 50 for state anxiety and 35 for trait anxiety. The most recent value is the individual's anxiety score. A high score indicates a high anxiety level, a small score indicates a low anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Ozcan, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No